CLINICAL TRIAL: NCT01490398
Title: Effect of Rosuvastatin on Coronary Flow Reserve in Hypertensive Patients
Brief Title: Rosuvastatin Effect on Serial Echocardiographic Measurement of Coronary Flow Velocity Reserve
Acronym: RESERVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0865
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension; Cardiovascular Risk Factors
Keywords: Hypertension; Rosuvastatin; Coronary flow reserve
MeSH Terms: conditions — Hypertension | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin (Experimental): Rosuvastatin 10mg qd for 12 months.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — After baseline assessment, the starting dose of rosuvastatin 10 mg will be given to study patients. If tolerated and LDL-C is > 100mg/dL after 2-4 weeks, the dose will be increased to 20 mg. Rosuvastatin treatment is scheduled to continue for 1 year without no further dose titration, and each patient will be followed at 2 months, 6 months and 1 year.
  Other Names: Crestor

SUMMARY:
In ASCOT study, lipid lowering with a statin provided additional beneficial effects in hypertensive patients with average levels of serum total cholesterol. However, the underlying mechanism of statins to improve clinical outcomes in hypertension is unclear and the effect of statins on coronary flow reserve (CFR) has not been examined in hypertensive patients. Therefore, it is clinically important and timely project to measure CFR non-invasively using echocardiography and to elucidate the mechanism of clinical benefits of statins in hypertensive patients with cardiovascular risk. The investigators try to evaluate the effect of rosuvastatin on CFR by measuring the change of CFR after 1 year treatment of rosuvastatin, and to correlate CFR with LDL-cholesterol and CRP.

DETAILED DESCRIPTION:
In hypertensive patients with high risk, lipid lowering with a statin provided additional beneficial effects in hypertensive patients with average levels of serum total cholesterol. However, the underlying mechanism of statins to improve clinical outcomes in hypertension is unclear. In patients with hypercholesterolemia or coronary atherosclerosis, several studies reported that level of LDL-cholesterol was inversely correlated with coronary blood flow reserve and suggested that statin improved coronary blood flow. Although it is speculated that statin may improve coronary blood flow by decreasing LDL cholesterol level and stabilizing atherosclerotic plaque in coronary atherosclerosis, the effect of statins on coronary flow reserve (CFR) has not been examined in hypertensive patients.

LDL cholesterol is expected to significantly decrease when rosuvastatin 20mg is administered. In addition to LDL-cholesterol lowering effect, the stabilization of atherosclerotic plaque and the regression of atheroma are observed during rosuvastatin treatment. Because of these beneficial effects of rosuvastatin, it may be expected that rosuvastatin will improve coronary blood flow even in hypertensive patients without hypercholesterolemia and the efficacy of rosuvastatin on CFR needs to be investigated in hypertensive patients with cardiovascular risk.

Morphologic assessment for the measurement of coronary lumen in the invasive coronary angiography is used as a gold standard to assess the stenosis in coronary diseases. However, as decrease of myocardial blood flow due to coronary artery disease could not be exactly evaluated by morphologic stenosis, the functional test was required to assess the significance of coronary artery stenosis, and CFR could be directly measured using Doppler guide wire since mid-1990s. Since the pathophysiological implication of coronary stenosis can be assessed using CFR measurement, CFR value is widely used in clinical practice as a very useful indicator to assess coronary stenosis severity in performing percutaneous coronary intervention. As a high frequency transducer with excellent resolution has been used, coronary artery can be directly imaged, and coronary flow velocity can be measured using echo-Doppler technique. As a result, CFR is easily measured in an echocardiography lab which could be measured only in a cardiac catheterization lab using Doppler guide wire in the past. It was confirmed that CFR values obtained by Doppler technique were same as those invasively obtained in a cardiac catheterization lab. The clinical usefulness and accuracy of the technique have been verified also in the diagnosis of coronary artery disease.

Therefore, it is clinically important and timely project to measure CFR non-invasively using echocardiography and to elucidate the mechanism of clinical benefits of statins in hypertensive patients with cardiovascular risk. We try to evaluate the effect of rosuvastatin on CFR by measuring the change of CFR after 1 year treatment of rosuvastatin, and to correlate CFR with LDL-cholesterol and CRP.

ELIGIBILITY:
Inclusion Criteria:

* Controlled Hypertension: treated SBP < 140 mmHg and DBP < 90 mmHg
* LDL cholesterol > 130 mg/dL
* Patients with statin-naive state, defined as receiving no statin therapy for more than 3 months during the previous 12 months
* Any 1 of these cardiovascular risk factors required: smoking, Type 2 DM, age over 55 (men) or 65 (women), peripheral vascular disease, history of cerebrovascular event, family history of early CHD before age 55, HDL cholesterol < 40 mg/dL

Exclusion Criteria:

* A previous history of intolerance or hypersensitivity to statins
* Uncontrolled hypertension; SBP ≥ 140 mmHg or DBP ≥ 90 mmHg
* Previous MI or currently treated angina pectoris
* Stroke, Transient ischemic attack < 3 months
* Secondary hypertension
* Fasting serum triglyceride > 500 mg/dL
* Clinical congestive heart failure
* Uncontrolled arrhythmia
* Left ventricular hypertrophy: LV mass index > 134g/m2 (male) or >110g/m2 (female)
* Concomitant clinically important respiratory, hematological, gastrointestinal, hepatic, renal or other disease
* Pregnant or lactating women and those of child-bearing potential

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change of coronary flow velocity reserve | 12 months
  Change of coronary flow velocity reserve from baseline to 1 year follow-up. For each patient, the averaged value of coronary flow velocity reserve will be obtained at baseline and 1 year follow-up.

SECONDARY OUTCOMES:
Change of averaged peak diastolic velocity | 12 months
  Change of averaged peak diastolic velocity from baseline to study end.
Change of CRP | 12 months
  Change of CRP from baseline to study end.
Change of LDL cholesterol | 12 months
  Change of LDL cholesterol from baseline to study end.

CONTACTS AND LOCATIONS:
Overall Officials: Duk Hyun Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Sun BJ, Hwang E, Jang JY, Kim DH, Song JM, Kang DH. Effect of rosuvastatin on coronary flow reserve in patients with systemic hypertension. Am J Cardiol. 2014 Oct 15;114(8):1234-7. doi: 10.1016/j.amjcard.2014.07.046. Epub 2014 Jul 30. PMID 25159238